CLINICAL TRIAL: NCT02536365
Title: Sensory Integration Therapy in Autism: Mechanisms and Effectiveness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: Thomas Jefferson University (Other); Queens College, The City University of New York (Other); Children's Specialized Hospital (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Sophie Molholm, Associate Professor, Albert Einstein College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2014-3795; R01HD082814 (NIH)
Record Dates: First submitted 2015-08-27; First posted 2015-08-31 (Estimated); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Autism
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Sensory Integration Therapy (Experimental): Children receive manualized SIT intervention that follows principles of sensory integration. SIT directly addresses the specific sensory factors hypothesized to underlie the child's functional skills difficulties and follows the Data Driven Decision Making Process, to tailor the intervention to the child's specific sensory issues.
  Interventions: Behavioral: Sensory Integration Therapy
- Applied Behavioral Analysis (Active Comparator): This involves examination of environmental variables that influence behavior and altering those variables to improve the child's skills. Intervention is individualized based on identified needs of the child, assessment of environmental variables impacting their performance of specific functional skills, and their abilities.
  Interventions: Behavioral: Applied Behavioral Analysis
- No Treatment (No Intervention): Treatment as usual will occur through the treatment period. As with the other treatment conditions, the participant agrees to refrain from beginning new treatments during participation in this study.

INTERVENTIONS:
Behavioral: Sensory Integration Therapy — Children in the SIT treatment group will receive a manualized SIT intervention that follows the principles of sensory integration.
  Arms: Sensory Integration Therapy
Behavioral: Applied Behavioral Analysis — Children in the ABA treatment group will receive intervention that follows the principles of Applied Behavioral Analysis.
  Arms: Applied Behavioral Analysis

SUMMARY:
A common feature of ASD is over or under sensitivity to the environment and difficulty putting sensory information together in an orderly way, referred to here as sensory issues. Building on previous work, this study will test the efficacy of Sensory Integration Therapy (SIT), a non-invasive intervention to improve functional skills in children with ASD, in comparison to commonly applied ABA behavioral treatments, in the treatment of ASD symptoms. A total of 180 children with ASD and sensory issues in the greater New York City Metropolitan area will complete this study.

DETAILED DESCRIPTION:
Autism Spectrum Disorders (ASD) are among the most common neurodevelopmental disorder with estimated costs of treatment across the lifespan of $3.2 million. A common feature of ASD is over or under sensitivity to the environment and difficulty putting sensory information together in an orderly way, referred to here as sensory issues. Such sensory issues are now included in the diagnostic criteria in the DSM5 under the Restrictive and Repetitive Behaviors and Interests Criteria. These sensory issues have a deleterious effect on functional skills and limit participation in work, education, and social activities for individuals with ASD and their family. Building on previous work, this study seeks to extend understanding of Sensory Integration Therapy (SIT) as a non-invasive intervention to improve functional skills in children with ASD and sensory issues, and to test its efficacy in comparison to commonly used applied behavioral treatments. Further, the investigators will explore the proposed neurobiological mechanisms by which this intervention may work, and phenotypic moderators of outcome. This study utilizes a randomized trial to compare SIT to a commonly used behavioral intervention to evaluate outcomes on functional skills as a basis for improved independence over the lifetime. A total of 180 children with ASD and sensory issues in the greater New York City Metropolitan area will complete this study.

ELIGIBILITY:
Inclusion Criteria:

1. Between the ages of 6.0 and 9.5 at the time of enrollment
2. Have a diagnosis of ASD that is confirmed by our research certified licensed psychologist based on clinical impression, DSM-5 criteria, and cut off scores from the Autism Diagnostic Schedule -2 (ADOS) (or CARS; an adjustment made as a consequence of pandemic) and the Autism Diagnostic Interview - Revised (ADI-R)
3. Has a non-verbal cognitive level of 70 or above (IQ cutoff is based on feasibility study data, and we make exceptions on a case-by-case basis to as low as 65)
4. Demonstrate difficulty processing and integrating sensory information as measured by the Sensory Profile (SP; 3 or more subscales or total test score in the definite difference range; or the Sensory Integration and Praxis Test -SIPT-; score of -1.0 on 3 or more subtests)
5. Guardians willing to attend 3 weekly sessions for the duration of the period and to refrain from initiation of any new behavioral, therapeutic or alternative treatments during the study period
6. If on psychotropic medication, they are at a point where dosage and treatment are stabilized for the duration of the study.

Exclusion Criteria:

* Children who are receiving > 12 hours/week of ongoing ASD-related services(excluding their educational programing), or who are receiving more than one hour per week of services that closely approximate the experimental intervention, will be excluded. Additionally, for safety reasons, children with significant medical co-morbidities (e.g., major heart problems, blindness, deafness, cerebral palsy, Fragile X or Down Syndrome, or tuberous sclerosis) will not be allowed to participate.

Ages: 6 Years to 114 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 135 (Actual)
Dates: Start 2015-09; Primary Completion 2022-10-15 (Actual); Study Completion 2022-10-15 (Actual)

PRIMARY OUTCOMES:
The Pediatric Evaluation of Disability Inventory-Computer Adaptive Test (PEDI-CAT) Daily Living | Increase between week 0 and week 12 in functional adaptivity as assessed by PEDI-CAT, with follow up for stability of change at week 24
  The PEDI-CAT provides a valid and reliable assessment of the child's ability to perform daily living skills. The psychometric properties including validity and reliability are well documented and the PEDI-CAT showed good discriminant validity between groups of children with and without disabilities in all domains. Score estimates were found to be stable over time with strong test-retest reliability
The Assessment of Motor and Process Skills (AMPS) | Increase between week 0 and week 12 in functional adaptivity as assessed by AMPS, with follow up for stability of change at week 24
  An observation-based, standardized performance assessment of daily living skills . It has been standardized on more than 150,000 persons, ages 2-100 years of age, internationally and cross-culturally.

SECONDARY OUTCOMES:
Repetitive Behavior Scale-Revised (RBS-R) | Reduction between week 0 and week 12 in repetitive behavior scale score as assessed by RBS-R, with follow up for stability of change at week 24
  The RRB is a 43-item parent rating scale that measures the presence and severity of 6 types of repetitive behaviors: rituals/sameness (12 items), self-injurious behavior (8 items), stereotypic behavior (9 items), compulsive behavior (6 items), and restricted interests (3 items). The RBS-R yields an overall Total Score and six Subscale Scores, and has demonstrated reliability, stability, and validity in large autism samples.

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Molholm, Ph.D., Principal Investigator — Principal Investigator
Locations (1):
- Children's Specialized Hospital, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No
We will not be sharing IPD

REFERENCES:
- [Derived] Schaaf RC, Ridgway EM, Jones EA, Dumont RL, Foxe J, Conly T, Sancimino C, Yi M, Mailloux Z, Hunt JM, Kirschner L, Leiby BE, Molholm S. A Comparative Trial of Occupational Therapy Using Ayres Sensory Integration and Applied Behavior Analysis Interventions for Autistic Children. Autism Res. 2025 Oct;18(10):2120-2134. doi: 10.1002/aur.70099. Epub 2025 Aug 15. PMID 40815044